CLINICAL TRIAL: NCT04084873
Title: Emotional Regulation Brief Procedure for Fibromyalgia, Through the Internet
Brief Title: An Emotional Regulation Brief Procedure (PbRE) for Fibromyalgia Using ICT's
Acronym: PbRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: iTCC55
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Fibromyalgia; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental PBrE (Experimental): Participants are exposed to several words of emotional contents (positive, and negative). The differences between these words will allow the regulation and counter regulation of emotional processes (Schwager y Rothermund, 2013). The words are related to clinical and personal characteristics of the patients and they will promote an emotional identification that improve the emotional regulation (Kashdan, Barret y McKnight, 2015).
  Interventions: Behavioral: PBrE
- Control PBrE (Placebo Comparator): Participants are exposed to several neutral words. These words do not have any emotional content and there are no reasons to think that they have any effect over the emotional regulation.
  Interventions: Behavioral: PBrE-Control
- Control (Other): Participants do not receive the intervention.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: PBrE — PbRE is a word reading task implementing through an App developed for smartphones. The patient will choose emotional positive and negative words related to personal and clinical characteristics.
  Arms: Experimental PBrE
Behavioral: PBrE-Control — Participants are exposed to several neutral words. These words do not have any emotional content and there are no reasons to think that they have any effect over the emotional regulation.
  Arms: Control PBrE
Behavioral: Control — Participants do not receive the intervention.
  Arms: Control

SUMMARY:
The study aims is to test the efficacy of an emotional regulation procedure for fibromyalgia patients using Information and Communications Technologies (ICTs). This procedure is based in a task that implies exposition to emotional words. The principal hypothesis is that exposition will improve the clinical symptomatology because the procedure restore an adequate emotional regulation.

DETAILED DESCRIPTION:
Previous studies have demonstrated that FM patients have difficulties to process emotional words when they are compared to normal subjects (Mercado et al., 2013). This dysfunctional emotion regulation could show attentional bias and it could be a way to increase FM symptomatology as pain, and fatigue (Duscheck et al., 2014).

The emotion generation and its regulation through an experimental task as reading words is a well stablished procedure (Lang, Bradley y Cuthbert, 1997). This paradigm has been shown efficacy in clinical context, to reduce anxiety in social phobia (Masia et al., 1999; Baños, Quero y Botella, 2008), generalized anxiety disorders (Fracalanza, Kroner y Antony, 2014), personality disorders (Arntz et al., 2012), and depression (Chuang et al., 2016). To address the gap between the experimental results of this form of emotional regulation in FM patients, and its clinical application, the aim of this study is to evaluate the efficacy of a Brief Procedure of Emotional Regulation for Fibromyalgia (PbRE)

PbRE is a word reading task implementing through an App developed for smartphones. The patient will choose emotional positive and negative words related to personal and clinical characteristics. This exercise has been shown useful in analogous tasks in relational frame theory (Hussey y Barnes-Holmes (2012) or in bias computer training (Salemink et al., 2014).

ELIGIBILITY:
Inclusion Criteria:

* Met the American College of Rheumatology (ACR) 2010 research classification criteria for FM (Wolfe et al., 2010, 2011); as confirmed by a rheumatologist
* A minimum of 18 years of age
* Showed adequate reading comprehension
* Were able to use a smartphone
* Were able to sign an informed consent form.

Exclusion Criteria:

* Had any mental disorder treated by a psychiatrist
* Were scheduled for surgery in the next 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Combined Index of Severity in Fibromyalgia (ICAF). Change is being assessed | Through study completion, an average of 1 year
  The Combined Index of Severity in Fibromyalgia (ICAF) is a questionnaire that allows the classification of patients by severity in clinical practice. This analysis is a self-report questionnaire of 59 items constructed with the most common clinical manifestations of FM (Vallejo, Rivera, & Esteve-Vives, 2010). The ICAF questionnaire offers total scores, where higher scores indicate a more severe disease. This questionnaire also provides four factors: emotional, physical (pain, fatigue, sleep quality and functional capacity), active coping, and passive coping. Similar to the total score, higher scores on each factor indicate greater severity, with the exception of the active coping factor, where higher scores indicate a better way to cope with the disease.
Fibromyalgia Impact Questionnaire (FIQ). Change is being assessed | Through study completion, an average of 1 year
  The Fibromyalgia Impact Questionnaire (FIQ) (Burckhardt, Clark, & Bennett, 1991; Rivera & González, 2004) is a self-report questionnaire designed to evaluate the impact of the FM on the life of the patient. This 10-item questionnaire is widely used and covers the principal areas of interest, including physical functioning, pain, sleep, mental health, and fatigue. The score ranges from 0 to 100, where higher scores indicate a more severe impact of the disease.

SECONDARY OUTCOMES:
EuroQol-5D-5L | Through treatment completion, an average of 6 weeks
  The EuroQol-5D-L questionnaire (Herdman et al., 2011) is divided into 2 sections. The first section contains 5 questions about mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Five levels for answering are included (no problems, slight problems, moderate problems, severe problems and extreme problems), ranging from 1 to 5. The second part is a VAS score, which records the responder's self-evaluated health, where 0 is worst imaginable health and 100 is best imaginable health.
Credibility and Expectancy Questionnaire (CEQ) | Through treatment completion, an average of 6 weeks
  Patients' expectancy of treatment will be assessed with the Credibility and Expectancy Questionnaire (CEQ) (Devilly and Borkovec, 2010). Both factors (credibility and expectancy) have been shown to be stable across different populations with high internal consistency within each factor. The scale consists of six questions, with answer options rated on a 10-point scale and on a 1-100 % scale.
Client Satisfaction Questionnaire | Through treatment completion, an average of 6 weeks
  The Client Satisfaction Questionnaire, in its 8-item version (CSQ-8; Larsen et al. 1979), has been used most commonly to assess satisfaction in mental health services. This tool includes a brief standardized scale with good psychometric properties that provides an overall assessment of satisfaction. We used the Spanish version of the CSQ-8 (Vázquez et al., 2017).
Pain Catastrophizing Scale (PCS) | Through study completion, an average of 1 year
  The Pain Catastrophizing Scale (PCS) (Sullivan, Bishop, & Pivik, 1995) is a 13-item scale used to assess pain catastrophizing. Participants rated the frequency of 13 negative pain-related thoughts and feelings on a 5-point Likert scale from 0 (not at all) to 4 (all the time). The range of scores is 0 to 54. Higher scores indicate greater catastrophizing. We used the Spanish version of the PCS (García Campayo et al., 2008).
Acceptance and Action Questionnaire - II | Through study completion, an average of 1 year
  Acceptance and Action Questionnaire - II (Bond et al., 2011; Ruiz, et al., 2013). The AAQ-II is a general measure of experiential avoidance and psychological inflexibility. It consists of 7 items which are responded to by using a 7-point Likert scale. The items reflect an unwillingness to experience unwanted emotions and thoughts.
Short Form 12 Health Survey | Through study completion, an average of 1 year
  The Short Form 12 Health Survey (SF-12) (Vilagut et al., 2008; Ware & Keller, 1996) is a generic instrument used to assess health-related quality of life. It is a self-report survey of 12 items grouped into eight dimensions: physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role and mental health. The score ranges from 0 to 100 for every scale, where higher scores indicate better health.
Emotion Regulation Questionnaire | Through study completion, an average of 1 year
  The Emotion Regulation Questionnaire (Gross & John, 2003; Cabello, Salgero, Fernández-Berrocal & Gross, 2013) consist of 10 items which are responded to by using a 7-point Likert scale. The items are grouped into two dimensions: cognitive reappraisal and expressive suppression.

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel A. Vallejo, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arntz A, Hawke LD, Bamelis L, Spinhoven P, Molendijk ML. Changes in natural language use as an indicator of psychotherapeutic change in personality disorders. Behav Res Ther. 2012 Mar;50(3):191-202. doi: 10.1016/j.brat.2011.12.007. Epub 2012 Jan 4. PMID 22317755
- [Background] Bennett MP, Meulders A, Baeyens F, Vlaeyen JW. Words putting pain in motion: the generalization of pain-related fear within an artificial stimulus category. Front Psychol. 2015 Apr 30;6:520. doi: 10.3389/fpsyg.2015.00520. eCollection 2015. PMID 25983704
- [Background] Duschek S, Werner NS, Limbert N, Winkelmann A, Montoya P. Attentional bias toward negative information in patients with fibromyalgia syndrome. Pain Med. 2014 Apr;15(4):603-12. doi: 10.1111/pme.12360. Epub 2014 Jan 21. PMID 24447855
- [Background] Mercado F, Gonzalez JL, Barjola P, Fernandez-Sanchez M, Lopez-Lopez A, Alonso M, Gomez-Esquer F. Brain correlates of cognitive inhibition in fibromyalgia: emotional intrusion of symptom-related words. Int J Psychophysiol. 2013 May;88(2):182-92. doi: 10.1016/j.ijpsycho.2013.03.017. Epub 2013 Apr 2. PMID 23557844
- [Background] Montoya P, Sitges C, Garcia-Herrera M, Izquierdo R, Truyols M, Blay N, Collado D. Abnormal affective modulation of somatosensory brain processing among patients with fibromyalgia. Psychosom Med. 2005 Nov-Dec;67(6):957-63. doi: 10.1097/01.psy.0000188401.55394.18. PMID 16314601
- [Background] Schwager S, Rothermund K. Counter-regulation triggered by emotions: positive/negative affective states elicit opposite valence biases in affective processing. Cogn Emot. 2013;27(5):839-55. doi: 10.1080/02699931.2012.750599. Epub 2012 Dec 14. PMID 23237331